CLINICAL TRIAL: NCT07041736
Title: A Randomized Controlled Trial Evaluating Postoperative Pain and Antibacterial Effect of Ultrasonic and 980 nm Diode Laser Combination
Brief Title: Evaluating Postoperative Pain and Antibacterial Effect of Ultrasonic and 980 nm Diode Laser Combination
Acronym: Postoperative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Sabah Morad Sobhy, Healthcare and research, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-PD-25-12
Record Dates: First submitted 2025-06-13; First posted 2025-06-27 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Lasers, Semiconductor; Ultrasonography

STUDY DESIGN:
Intervention Model Description: this randomized controlled clinical trial included 120 patients that have single rooted teeth with necrotic pulp and periapical radioluceny. Patients were randomly assigned to receive root canal disinfection using either conventional techniquediode laser, ultrasonic irrigation, or a combination of both.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group I (conventional group) (Experimental): Access cavity preparation will be performed under strict aseptic condition and rubber dam isolation. Orifice location will be identified then, microbiological sample (S1) will be taken. The working length will be determined using an electronic apex locator (EAL) and will be confirmed using periapical radiograph. Root canal preparation will be performed using EdgeFile X7 nickel-titanium rotary system ((Edge Endo, Albuquerque, New Mexico, USA) driven by EndoEst motor mini (Geosoft Dent., Russia) endomotor till #40 taper 0.04 file in continuous rotation at 300 rpm and 2 Ncm.
  Interventions: Other: conventional irrigation
- Group II (Diode laser group) (Experimental): The same steps as mentioned in group I up to the use of saline solution for final irrigation. Then, the canal will be irradiated with 980 nm diode laser with optical fiber 200 µm (Lite medics, Italy) and power setting 1.2 watt in pulsed mode. The irradiation protocol will be a 5 sec. irradiation followed by a 10 sec. rest, which constituted one lasing cycle. The lasing cycle will be performed four times for each tooth. Microbiological sample (S2) will be taken after laser application.
  Interventions: Device: diode laser
- Group III (Ultrasonic group) (Experimental): The same as in group I however, during cleaning and shaping ProUltra PiezoFlow (Dentsply Tulsa Dental Specialties, Tulsa, OK, USA.) will be used for activation of the irrigating solution according to the manufacturer's recommendations. The needle will be operated using Satelec P5 Piezoelectric Ultrasonic Unit (Acteon, Mount Laurel, NJ, USA.) at power setting of 5. The stopper on the PiezoFlow needle will be set 1 mm short of binding in the canals, but not more than 75% of the WL. A syringe containing 5 mL of 2.5% NaOCl will be attached to the Piezoflow activation needle and the inactive needle will be inserted in the canal, and irrigant flow will be started before activation. During activation, the needle will be moved up and down passively in the canal (26). 5 ml of 17% EDTA (Colgate Oral Care Company, Waverly, Australia) for 1 min will be used for smear layer removal. 5 ml of saline solution will be used for final irrigation of the root canal to neutralize all the previously used
  Interventions: Device: Ultrasonic
- Group IV Ultrasonic+Diode (Experimental): The same steps as in group III then, 980 nm diode laser irradiation will be applied as in Group II and microbiological sample (S2) will be taken after laser application
  Interventions: Device: Diode laser; Device: Ultrasonic

INTERVENTIONS:
Device: diode laser — 980 nm diode laser with optical fiber 200 µm (Lite medics, Italy) and power setting 1.2 watt in pulsed mode. The irradiation protocol will be a 5 sec. irradiation followed by a 10 sec. rest, which constituted one lasing cycle. The lasing cycle will be performed four times for each tooth.
  Arms: Group II (Diode laser group)
Other: conventional irrigation — After each file use, the root canal will be irrigated with 5ml of freshly prepared 2.5% sodium hypochlorite (NaOCl) solution (Alex. Deteregents and Chemical Co., Egypt) for 1 minute using a 31-gauge Navi-Tip flexible irrigating needle (Navi-Tip, Ultradent product, South Jourdan, UT). 5 ml of 17% EDTA (Colgate Oral Care Company, Waverly, Australia) for 1 min will be used for smear layer removal. 5 ml of saline solutio
  Arms: Group I (conventional group)
Device: Diode laser — 980 nm diode laser with optical fiber 200 µm (Lite medics, Italy) and power setting 1.2 watt in pulsed mode. The irradiation protocol will be a 5 sec. irradiation followed by a 10 sec. rest, which constituted one lasing cycle. The lasing cycle will be performed four times for each tooth.
  Arms: Group IV Ultrasonic+Diode
Device: Ultrasonic — The needle will be operated using Satelec P5 Piezoelectric Ultrasonic Unit (Acteon, Mount Laurel, NJ, USA.) at power setting of 5. The stopper on the PiezoFlow needle will be set 1 mm short of binding in the canals, but not more than 75% of the WL. A syringe containing 5 mL of 2.5% NaOCl will be attached to the Piezoflow activation needle and the inactive needle will be inserted in the canal, and irrigant flow will be started before activation. During activation, the needle will be moved up and down passively in the canal
  Arms: Group III (Ultrasonic group); Group IV Ultrasonic+Diode

SUMMARY:
This study is a parallel randomized controlled clinical trial that was designed and interpreted according to Preferred Reporting Items for Randomized Trial in Endodontics (PRIRATE) 2020 guidelines. Patients of age range between 20 and 35 years old from the outpatient clinic of Endodontic Department, Faculty of Dental Medicine for Girls, Al-Azhar University will participate in this study. These patients have single rooted teeth with necrotic pulp and periapical radiolucency. Patients will be informed about all the study's procedures. They will be included in the study after fulfilling the inclusion criteria and sign an informed consent.Inclusion Criteria:

* Patients have mature teeth with closed apex.
* Single rooted teeth with root canal form type I.
* Asymptomatic.
* Have Periapical radiolucency with diameter up to 5 mm.
* Restorable teeth.

Exclusion Criteria:

* Patients with symptomatic apical periodontitis.
* Systemic disease.
* Physical or mental disability.
* Root fracture and tooth mobility.

DETAILED DESCRIPTION:
Ethical approval for the human study was obtained by the Research Ethics Committee (REC) of the Faculty of Dental Medicine for Girls, Al-Azhar University, Egypt . All patients were provided with an informed consent form outlining the study's details including potential benefits and risks, which they read and signed prior to participation. Sample size calculation was performed using G*Power version 3.1.9.7 based on the results of a previous study . A power analysis was designed to have adequate power to apply a two-sided statistical test to reject the null hypothesis that there is no difference between groups. By adopting an alpha level of (0.05) and a beta of (0.2), i.e. power = 80% and an effect size (d) of (0,332) calculated based on the primary outcome (Postoperative pain) and the results of a previous study. The predicted sample size (n) was (104), i.e., 26 subjects per group. This number is increased to 30 subjects per group to compensate for a drop-out rate of 15%.

ELIGIBILITY:
Inclusion Criteria:

* Patients have mature teeth with closed apex.
* Single-rooted teeth with root canal form type I.
* Asymptomatic.
* Have periapical radiolucency with a diameter of up to 5 mm.
* Restorable teeth.

Exclusion Criteria:

* Patients with symptomatic apical periodontitis.
* Systemic disease.
* Physical or mental disability.
* Root fracture and tooth mobility.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-03 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain evaluation | after 24,48 and 72hours of the treatment
  Postoperative pain will be recorded using numerical rating scale (NRS) with minimum value 0 and maximum value 10 (worst pain).

SECONDARY OUTCOMES:
Microbiological analysis | 24,48 hours
  Microbiological analysis of samples (S1&S2) will be performed to evaluate the percentage of reduction in the number of Colony Forming Units (CFU) of aerobic and anaerobic bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Sabah M. Sobhy, PHD, Principal Investigator — Endodontic Department, Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egyp
Locations (1):
- from the outpatient clinic of Endodontic Department, Faculty of Dental Medicine for Girls, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dragana R, Jelena M, Jovan M, Biljana N, Dejan M. Antibacterial efficiency of adjuvant photodynamic therapy and high-power diode laser in the treatment of young permanent teeth with chronic periapical periodontitis. A prospective clinical study. Photodiagnosis Photodyn Ther. 2023 Mar;41:103129. doi: 10.1016/j.pdpdt.2022.103129. Epub 2022 Sep 23. PMID 36156313
- [Background] Ghonem Z A, Mustafa MH, Shishiny A. Antibacterial Efficacy of Diode laser 810nm on Enterococcus Faecalis on Primary Teeth, an invitro study. Al-Azhar Journal of Dentistry. 2024; 11: 32-8. doi.org/10.58675/2974-4164.1623.
- [Background] Nair PN. Pathogenesis of apical periodontitis and the causes of endodontic failures. Crit Rev Oral Biol Med. 2004 Nov 1;15(6):348-81. doi: 10.1177/154411130401500604. PMID 15574679
- [Background] Fahim SZ, Ghali RM, Hashem AA, Farid MM. The efficacy of 2780 nm Er,Cr;YSGG and 940 nm Diode Laser in root canal disinfection: A randomized clinical trial. Clin Oral Investig. 2024 Feb 26;28(3):175. doi: 10.1007/s00784-024-05563-z. PMID 38403667